CLINICAL TRIAL: NCT01007474
Title: One Hospital ClinicalService Project on Patients Implanted With Medtronic Implantable Devices or Treated by Medtronic Therapies
Brief Title: One Hospital ClinicalService Project
Acronym: OHCS
Status: Withdrawn | Type: Observational
Why Stopped: The One Hospital ClinicalService project involves the provision of services to hospitals, and is not a clinical study. As such, this service offering should not be listed on ClinicalTrials.gov.
Sponsor: Medtronic Italia (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT-OHCS
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Arrhythmias, Cardiac; Bradycardia; Syncope
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia; Syncope | interventions — Defibrillators, Implantable; Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Implantable Cardioverter-Defibrillator (ICD) — Medtronic market-released implantable cardioverter-defibrillator
Device: Implantable Pacemaker Generator (IPG) — Medtronic market-released implantable pacemaker generator
Device: Implantable Loop Recorder (ILR) — Medtronic market-released implantable loop recorder
Device: Cardiac Resynchronization Therapy-Defibrillator (CRT-D) — Medtronic market-released cardiac resynchronization therapy defibrillator
Device: Implantable devices working as neurostimulators, stents, spinal/bone devices or other applications — Medtronic market-released implantable devices used as neurostimulators, stents, spinal/bone devices or for other applications

SUMMARY:
The One Hospital ClinicalService Project is an integrated system composed by a network of International Hospital Departments, a clinical data repository and a shared environment for the collection, management, analysis and reporting of clinical and diagnostics data from patients treated by Medtronic therapies or patients wearing Medtronic implantable devices used within their intended use. The One Hospital ClinicalService is composed by a suite of systematic, data-guided activities designed to bring about immediate improvements in health delivery in particular settings. Data are prospectively collected. An independent committee of physicians prospectively identifies key clinical questions on a yearly basis for development of quality improvement activities, analyses and publications. A charter, approved by Hospital Istitutional Review Boards or other Hospital entities, assigns the ownership of data to the centers and governs the conduct of the project and the relationship of the scientific committee and Medtronic. Hospital is the data controller, while Medtronic is the data processor on behalf of the Hospital. Data collected for quality improvement purposes may be mined to perform clinical research.

DETAILED DESCRIPTION:
One Hospital ClinicalService is a project aiming to provide information and analysis of clinical and device data, back to the treating healthcare providers regarding their own patients, in order to help those healthcare providers improve outcomes and understanding of their patients' care or patients' management.

The mission of the One Hospital ClinicalService Project is to improve outcomes and comprehension of diagnostic and therapeutic strategies applied to patients wearing Medtronic implantable devices or treated by Medtronic therapies. One Hospital ClinicalService provides services to evaluate and improve the quality of clinical care in the International clinical practice.

One Hospital ClinicalService collects acute and chronic patient and device data in a large population during routine usage of the device, without specific study interventions, and always within the approved intended use of the device.

One Hospital ClinicalService uses a core database which can be expanded with specific data sets for particular patient populations, diseases, therapies, devices or features.

One Hospital ClinicalService, with its prospective data collection and its data management infrastructure, forms a data-bank where physicians collect patient data and from which they receive reports about clinical and device diagnostics data. Usage and understanding of diagnostics data may help physicians to optimize tailor device programming and patient therapies. This data-bank, queried by retrospective statistical analyses, may help physicians in quality improvement activities, education, research and scientific activities.

Some examples of scientific focus available through the One Hospital ClinicalService Project include:

* Describing the use of implantable devices, such as cardioverter defibrillator (ICD), pacemakers, implantable loop recorders or others in the Italian clinical practice
* Identifying predictors or clinical variables correlated with clinical outcomes or therapy response
* Evaluating and testing methods to optimize device programming and patient therapy via device diagnostics or patient reports

ELIGIBILITY:
Inclusion Criteria:

* Patients wearing a Medtronic market-released device or treated by a Medtronic therapy who have signed a patient data release and informed consent form

Exclusion Criteria:

* Patients unwilling or unable to cooperate or give voluntary consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients who received a Medtronic device or were treated by Medtronic therapy (currently available or future market-released devices) at one of the participating International Hospitals.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-01; Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | 10 years

SECONDARY OUTCOMES:
Hospitalizations | 10 years

OTHER OUTCOMES:
Device interventions | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Boriani, MD, Study Chair — Cardiology Department, Policlinico di Modena, University of Modena and Reggio Emilia
Locations (41):
- Stauferklinikum Mutlangen, Mutlangen, Germany
- Landspitali University Hospital, Reykjavik, Iceland
- India (2):
  - Eternal Hospital, Jaipur
  - Fortis Escort Heart Institute, New Delhi
- Italy (25):
  - S.Orsola Malpigli, Bologna
  - Ospedale Civile di Bolzano, Bolzano
  - A.O. S.Sebastiano di Caserta, Caserta
  - S. Anna Hospital, Como
  - A.O. Santa Croce e Carle, Cuneo
  - Ospedale Santa Croce, Fano
  - A.Ospedaliero Universitaria Careggi, Florence
  - Ospedali Riuniti Leonardi-Riboli, Lavagna
  - ASL 2 Avellino, Mercogliano
  - Istituto Auxologico Italiano, Milan
  - Istituto Ca' Granda-Niguarda, Milan
  - Ospedale Luigi Sacco, Milan
  - San Carlo Borromeo, Milan
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - A.O. di Parma, Parma
  - Policlinico S. Matteo, Pavia
  - A.O. San Salvatore di Pesaro, Pesaro
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Fatebenefratelli S:Giovalli Calibita, Roma
  - Policlinico A. Gemelli, Roma
  - San Filippo Neri Hospital, Roma
  - Istituto Clinico Humanitas, Rozzano
  - ASL Teramo, Teramo
  - A.O. S.Maria della Misericordia, Udine
  - Ospedale S. Maria della Misericordia, Urbino
- Japan (5):
  - Osaka University Hospital, Suita, Osaka
  - Tokyo Medical and Dental University Hospital, Bunkyō-Ku, Tokyo
  - Kagawa University Hospital, Kagawa
  - Saiseikai Kawaguchi General Hospital, Kawaguchi
  - Toyohashi Heart Center, Toyohashi
- Saudi Arabia (2):
  - King Fadh Atmnd Forces Hospital, Jeddah
  - Prince Sultan Cardiac Center, Riyadh
- Mediclinic Panorama Hospital, Cape Town, South Africa
- Hallandssjukhus Varberg, Varberg, Sweden
- United Kingdom (3):
  - Blackpool Victoria Hospital, Blackpool
  - Greater Glasgow Health Board, Glasgow
  - Central Manchester University Hospital NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Moltrasio M, Iacopino S, Arena G, Pieragnoli P, Molon G, Manfrin M, Verlato R, Ottaviano L, Rovaris G, Catanzariti D, Cipolletta L, Nicolis D, Cattafi G, Tondo C; 1STOP ClinicalService centers. First-line therapy: insights from a real-world analysis of cryoablation in patients with atrial fibrillation. J Cardiovasc Med (Hagerstown). 2021 Aug 1;22(8):618-623. doi: 10.2459/JCM.0000000000001176. PMID 34009837
- [Derived] Giannola G, Torcivia R, Airo Farulla R, Cipolla T. Outsourcing the Remote Management of Cardiac Implantable Electronic Devices: Medical Care Quality Improvement Project. JMIR Cardio. 2019 Dec 18;3(2):e9815. doi: 10.2196/cardio.9815. PMID 31845898
- [Derived] Ricciardi D, Arena G, Verlato R, Iacopino S, Pieragnoli P, Molon G, Manfrin M, Allocca G, Cattafi G, Sirico G, Rovaris G, Sciarra L, Nicolis D, Tondo C. Sex effect on efficacy of pulmonary vein cryoablation in patients with atrial fibrillation: data from the multicenter real-world 1STOP project. J Interv Card Electrophysiol. 2019 Oct;56(1):9-18. doi: 10.1007/s10840-019-00601-3. Epub 2019 Aug 26. PMID 31452001
- [Derived] Perego GB, Iacopino S, Molon G, Arena G, Verlato R, Pieragnoli P, Curnis A, Allocca G, Nicolis D, Sciarra L, Catanzariti D, Senatore G, Rovaris G, Brasca F, Tondo C; ClinicalService 1STOP project i Project Investigators. Cryoablation for paroxysmal and persistent AF in patients with structural heart disease and preserved ejection fraction: Clinical outcomes from 1STOP, a multicenter observational project. J Cardiol. 2019 Jul;74(1):19-26. doi: 10.1016/j.jjcc.2019.02.015. Epub 2019 Apr 1. PMID 30948185
- [Derived] Landolina M, Arena G, Iacopino S, Verlato R, Pieragnoli P, Curnis A, Lunati M, Rauhe W, Senatore G, Sciarra L, Molon G, Agricola PMG, Padeletti L, Tondo C. Center experience does not influence long-term outcome and peri-procedural complications after cryoballoon ablation of paroxysmal atrial fibrillation: Data on 860 patients from the real-world multicenter observational project. Int J Cardiol. 2018 Dec 1;272:130-136. doi: 10.1016/j.ijcard.2018.07.051. Epub 2018 Jul 18. PMID 30045822
- [Derived] Stabile G, Tondo C, Curnis A, Lunati M, Manfrin M, Molon G, Sciarra L, Mantica M, Iacopino S, Arena G, Landolina M, Arestia A, Verlato R. Efficacy of cryoballoon ablation in patients with paroxysmal atrial fibrillation without time to pulmonary vein isolation assessment. Int J Cardiol. 2018 Dec 1;272:118-122. doi: 10.1016/j.ijcard.2018.07.070. Epub 2018 Jul 20. PMID 30037629
- [Derived] Lunati M, Arena G, Iacopino S, Verlato R, Tondo C, Curnis A, Porcellini S, Sciarra L, Molon G, Senatore G, Leoni L, Perego GB, Rauhe W, Pepi P, Landolina M. Is the time between first diagnosis of paroxysmal atrial fibrillation and cryoballoon ablation a predictor of efficacy? J Cardiovasc Med (Hagerstown). 2018 Aug;19(8):446-452. doi: 10.2459/JCM.0000000000000688. PMID 29927782
- [Derived] Gasparini M, Kloppe A, Lunati M, Anselme F, Landolina M, Martinez-Ferrer JB, Proclemer A, Morani G, Biffi M, Ricci R, Rordorf R, Mangoni L, Manotta L, Grammatico A, Leyva F, Boriani G. Atrioventricular junction ablation in patients with atrial fibrillation treated with cardiac resynchronization therapy: positive impact on ventricular arrhythmias, implantable cardioverter-defibrillator therapies and hospitalizations. Eur J Heart Fail. 2018 Oct;20(10):1472-1481. doi: 10.1002/ejhf.1117. Epub 2017 Dec 18. PMID 29251799
- [Derived] Boriani G, Lip GYH, Ricci RP, Proclemer A, Landolina M, Lunati M, Padeletti L, Zanotto G, Molon G, Biffi M, Rordorf R, Quartieri F, Gasparini M. The increased risk of stroke/transient ischemic attack in women with a cardiac implantable electronic device is not associated with a higher atrial fibrillation burden. Europace. 2017 Nov 1;19(11):1767-1775. doi: 10.1093/europace/euw333. PMID 28031277
- [Derived] Padeletti L, Curnis A, Tondo C, Lunati M, Porcellini S, Verlato R, Sciarra L, Senatore G, Catanzariti D, Leoni L, Landolina M, Delise P, Iacopino S, Pieragnoli P, Arena G. Pulmonary Vein Isolation with the Cryoballoon Technique: Feasibility, Procedural Outcomes, and Adoption in the Real World: Data from One Shot Technologies TO Pulmonary Vein Isolation (1STOP) Project. Pacing Clin Electrophysiol. 2017 Jan;40(1):46-56. doi: 10.1111/pace.12975. Epub 2016 Dec 22. PMID 27862043
- [Derived] Zoppo F, Facchin D, Molon G, Zanotto G, Catanzariti D, Rossillo A, Baccillieri MS, Menard C, Comisso J, Gentili A, Grammatico A, Bertaglia E, Proclemer A. Improving atrial fibrillation detection in patients with implantable cardiac devices by means of a remote monitoring and management application. Pacing Clin Electrophysiol. 2014 Dec;37(12):1610-8. doi: 10.1111/pace.12474. Epub 2014 Aug 12. PMID 25113510
- [Derived] Ricci RP, Pignalberi C, Landolina M, Santini M, Lunati M, Boriani G, Proclemer A, Facchin D, Catanzariti D, Morani G, Gulizia M, Mangoni L, Grammatico A, Gasparini M; ClinicalService cardiological centres. Ventricular rate monitoring as a tool to predict and prevent atrial fibrillation-related inappropriate shocks in heart failure patients treated with cardiac resynchronisation therapy defibrillators. Heart. 2014 Jun;100(11):848-54. doi: 10.1136/heartjnl-2013-305259. Epub 2014 Mar 28. PMID 24682569
- [Derived] Verlato R, Facchin D, Catanzariti D, Molon G, Zanotto G, Morani G, Brieda M, Zanon F, Delise P, Leoni L, Comisso J, Campo C. Clinical outcomes in patients with implantable cardioverter defibrillators and Sprint Fidelis leads. Heart. 2013 Jun;99(11):799-804. doi: 10.1136/heartjnl-2012-303259. Epub 2013 Feb 22. PMID 23434626
- [Derived] Boriani G, Santini M, Lunati M, Gasparini M, Proclemer A, Landolina M, Padeletti L, Botto GL, Capucci A, Bianchi S, Biffi M, Ricci RP, Vimercati M, Grammatico A, Lip GY; Italian ClinicalService Project. Improving thromboprophylaxis using atrial fibrillation diagnostic capabilities in implantable cardioverter-defibrillators: the multicentre Italian ANGELS of AF Project. Circ Cardiovasc Qual Outcomes. 2012 Mar 1;5(2):182-8. doi: 10.1161/CIRCOUTCOMES.111.964205. Epub 2012 Feb 28. PMID 22373906
- [Derived] Landolina M, Gasparini M, Lunati M, Iacopino S, Boriani G, Bonanno C, Vado A, Proclemer A, Capucci A, Zucchiatti C, Valsecchi S, Ricci RP, Santini M; Cardiovascular Centers Participating in the ClinicalService Project. Long-term complications related to biventricular defibrillator implantation: rate of surgical revisions and impact on survival: insights from the Italian Clinical Service Database. Circulation. 2011 Jun 7;123(22):2526-35. doi: 10.1161/CIRCULATIONAHA.110.015024. Epub 2011 May 16. PMID 21576653
- [Derived] Santini M, Gasparini M, Landolina M, Lunati M, Proclemer A, Padeletti L, Catanzariti D, Molon G, Botto GL, La Rocca L, Grammatico A, Boriani G; cardiological centers participating in ClinicalService Project. Device-detected atrial tachyarrhythmias predict adverse outcome in real-world patients with implantable biventricular defibrillators. J Am Coll Cardiol. 2011 Jan 11;57(2):167-72. doi: 10.1016/j.jacc.2010.08.624. PMID 21211688